CLINICAL TRIAL: NCT04258384
Title: The Turkish Cross-Cultural Adaptation, Validity and Reliability of Vanderbilt Multidimensional Pain Coping Inventory
Brief Title: The Turkish Cross-Cultural Adaptation, Validity and Reliability of VMPCI
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: 37068608-6100-15-1685
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Pain, Chronic
Keywords: Rheumatoid Arthritis, pain, coping, validity, reliability
MeSH Terms: conditions — Chronic Pain; Arthritis, Rheumatoid; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: The study included individuals whose native language is Turkish, who are literate, over the age of 18, diagnosed with rheumatoid arthritis, without cognitive impairment and communication problems, and who want to participate in the study.
  Interventions: Other: survey application

INTERVENTIONS:
Other: survey application — Data collection tools used in the study; Demographic Data Form, Mcgill and Melzack Pain Questionnaire, Short Form-36 (SF-36), Vanderbilt Multidimensional Pain Coping Inventory (VMPCI), Pain Coping Inventory (PCI), Pain Coping Scale were used.

SUMMARY:
This study was planned to adapt the Vanderbilt Multidimensional Pain Coping Inventory into Turkish, to investigate its cultural adaptation, validity and reliability. The study was completed with 352 volunteers who fulfilled the criteria to be included in the Rheumatology Clinic of Istanbul Haydarpaşa Numune Training and Research Hospital. Data collection tools used in the study; Demographic Data Form, Mcgill and Melzack Pain Questionnaire, Short Form-36 (SF-36), Vanderbilt Multidimensional Pain Coping Inventory (VMPCI), Pain Coping Inventory (PCI), Pain Coping Scale were used.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, progressive, inflammatory, autoimmune disease of unknown etiology, mainly affecting synovial joints, causing loss of function. The main reason that directs RA patients to medical treatment is pain. Chronic pain causes limitation of movement, sleep problems, fatigue, stress and depression, as well as physiological and psychological problems that cause negative effects on the quality of life of the individual. The patient's thoughts, expectations, and methods of coping with pain are effective in pain control. In order to identify and treat the painful condition, individual coping methods of the patient and the effectiveness of these methods should be evaluated. This study was planned to adapt the Vanderbilt Multidimensional Pain Coping Inventory into Turkish, to investigate its cultural adaptation, validity and reliability. The study was completed with 352 volunteers who fulfilled the criteria to be included in the Rheumatology Clinic of Istanbul Haydarpasa Numune Training and Research Hospital. Data collection tools used in the study; Demographic Data Form, Mcgill and Melzack Pain Questionnaire, Short Form-36 (SF-36), Vanderbilt Multidimensional Pain Coping Inventory (VMPCI), Pain Coping Inventory (PCI), Pain Coping Scale were used. The language validity of the Turkish form of the scale was provided by the translation-back translation method. Expert opinion was obtained for scale of validity. In order to evaluate the reliability of the Turkish version of the scale; internal consistency coefficient, test retest and parallel form methods were used. After all these analyzes, the reliability and validity of the Turkish version of the VMPCI scale was obtained. In addition to this study, the descriptive characteristics of the sample, SF-36 scale, Mcgill and Melzack Pain Questionnaire results were examined alone and together with the sub-dimensions of the scale.

ELIGIBILITY:
Inclusion Criteria:The study included individuals whose native language is Turkish, who are literate, over the age of 18, diagnosed with rheumatoid arthritis, without cognitive impairment and communication problems, and who want to participate in the study.

-

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included individuals whose native language is Turkish, who are literate, over the age of 18, diagnosed with rheumatoid arthritis, without cognitive impairment and communication problems, and who want to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Vanderbilt Multidimensiyonel Pain Coping Inventory | 15 minutes
  Patients are asked to mark their preferred behaviors and the thoughts of the hospital when their pain is moderate or high intensity.

SECONDARY OUTCOMES:
Demographic Data Form | 5 minutes
  This form prepared by the researcher includes the socio-demographic characteristics of the patients who will participate in the study, the history of the disease, findings related to the characteristics related to pain and exacerbations.
SF36 | 10 minutes
  The scale includes 36 questions that evaluate 8 sub-scales of health as physical function, physical role difficulty, pain, general health, vitality, social function, emotional role function, mental health topics.
McGill Melzack Pain Questionnaire | 5 minutes
  It consists of four parts. In the first part, it is desired to mark the shape of the pain on the figure and use the letters "D" if deep pain is heard, "Y" if the pain is superficial, and "D - Y" if the two conditions are experienced at the same time. In the second part, there are twenty word groups that define pain in terms of sensory, perceptual and evaluation. Each of the word groups consists of two-six words that describe pain in different ways. In the third part, there is a time relationship of pain. It includes phrases to understand the continuity and frequency of pain and to identify situations that increase or decrease pain. The last section contains words that indicate the severity of pain. With this questionnaire used in the study, it was aimed to determine the location of the pain, the feeling of the patient, the relationship of pain time, the severity of the pain and the level of livable pain for the patient.
Pain Coping Scale | 5 minutes
  The scale determines how chronic pain patients cope with organic or psychogenic pain. It consists of self-coping, helplessness, conscious cognitive interventions, and medical remedy sub-scales.
Pain Coping Inventory | 5 minutes
  It evaluates how often patients with chronic pain use behavioral and cognitive methods to deal with pain. Active as transforming pain, moving away and reducing demand; There are six passive sub-dimensions as retreat, anxiety and rest.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Gelisim University, Istanbul, Istanbul/ Avcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No